CLINICAL TRIAL: NCT01260194
Title: An Open-label, Multicentre Phase IV Study of Trastuzumab in Combination With the Standard Therapy (as Per Routine Clinical Practice) as First-line Therapy in Patients With HER2 Positive Metastatic Gastric Cancer
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With Standard Chemotherapy in Patients With HER Positive Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25477
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: trastuzumab [Herceptin] — Loading dose of 8 mg/kg on day 1, followed by 6 mg/kg intravenous infusion every 3 weeks until disease progression in combination with standard chemotherapy

SUMMARY:
This open-label, multi-center study will evaluate the efficacy and safety of Herceptin (trastuzumab) in combination with standard chemotherapy as first-line treatment in patients with HER2 positive metastatic adenocarcinoma of the stomach or gastro-esophageal junction. Patients will receive standard chemotherapy for a maximum of 6 cycles, and 8 mg/kg Herceptin as loading dose on day 1, followed by 6 mg/kg intravenous infusion every 3 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Histologically confirmed adenocarcinoma of the stomach or gastro-esophageal junction with advanced or metastatic disease, not amenable to curative therapy
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* HER2 positive tumor (primary tumor or metastasis
* ECOG Performance status 0, 1 or 2
* Life expectancy of at least 3 months

Exclusion Criteria:

* Previous chemotherapy for advanced or metastatic disease less than 6 month before study start
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (patients with partial or total gastrectomy are allowed to participate in the study)
* Patients with active (significant or uncontrolled) gastrointestinal bleeding
* Residual relevant toxicity resulting from previous chemotherapy
* Other malignancy within the last 5 years (except carcinoma in situ of the cervix, or basal cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- India (6):
  - Bangalore, Karnataka
  - New Delhi, National Capital Territory of Delhi
  - Bangalore
  - Nagpur
  - Noida
  - Vishakpatnam

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab: Trastuzumab was administered at a loading dose of 8 milligram per kilogram (mg/kg) body weight on Day 1, followed by 6 mg/kg intravenous infusion every 3 weeks plus standard chemotherapy as per Investigator's discretion or as per institutional practice, until disease progression, early withdrawal due to unmanageable toxicity, or consent withdrawal.
Period: Overall Study
Arm/Group | Trastuzumab
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal of Consent | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug and did not report any major protocol violation.
Groups:
- Trastuzumab: Trastuzumab was administered at a loading dose of 8 mg/kg on Day 1, followed by 6 mg/kg intravenous infusion every 3 weeks plus standard chemotherapy as per Investigator's discretion or as per institutional practice, until disease progression, early withdrawal due to unmanageable toxicity, or consent withdrawal.
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.27)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: The PFS was defined as the median time between the day of enrollment and the first documentation of progressive disease (PD) or date of death, whichever occurred first. PD was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeters [mm]) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. The censoring date was the last date of "last tumor measurement," "last date of study drug treatment," or "last follow-up." The median PFS time with 95% confidence interval (CI) was estimated using Kaplan Meier method.
Time Frame: Baseline up to PD or death (maximum up to 22 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
days | 254.0 [52.0 to 508.0]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of enrollment to the date of the death (from any cause). If no death was observed, censored observations were taken into account in the analysis. The censoring date was the last date of "last tumor measurement," "last date in drug log," or "last follow-up." The median overall survival time with 95% CI was estimated using Kaplan Meier method.
Time Frame: Baseline up to death (maximum up to 22 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
days | 508.0 [82.0 to NA] — Data could not be estimated due to insufficient number of deaths (less than or equal to [<=] 50% participants).

3. Secondary Outcome: Percentage of Participants With Overall Tumor Response
Description: Overall tumor response was defined as the occurrence of either a confirmed complete response (CR) or a partial response (PR) as best overall response as determined by the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version (v) 1.1 from confirmed radio-graphic evaluations of target and non-target lesions. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease; all nodes, both target and non-target, must decrease to normal (short axis less than [<]10 mm); no new lesions. PR was defined as greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions (the short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions); no unequivocal progression of non-target disease; no new lesions.
Time Frame: Baseline up to PD or death (maximum up to 22 months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
percentage of participants | 50 [9.4 to 99.2]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit Response (CBR)
Description: CBR was defined as any response among stable disease (SD) for 6 weeks or longer, CR, or PR as determined by the RECIST v 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease; all nodes, both target and non-target, must decrease to normal (short axis <10 mm); no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions (the short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions); no unequivocal progression of non-target disease; no new lesions. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. SD was defined as not qualifying for CR, PR, or PD.
Time Frame: Baseline up to PD or death (maximum up to 22 months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
percentage of participants | 75.0 [29.2 to 100.0]

5. Secondary Outcome: Duration of Response (DR)
Description: DR was based on RECIST criteria v1.1 and was defined as time from date the CR or PR was first recorded to the date on which PD was first noted. CR: complete disappearance of all target lesions and non-target disease, with the exception of nodal disease; all nodes, both target and non-target, must decrease to normal (short axis <10 mm); no new lesions. PR: >=30% decrease under baseline of the sum of diameters of all target lesions; no unequivocal progression of non-target disease; no new lesions. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions and/or appearance of 1 or more new lesions. For the participants with no documented progression after CR or PR, the censored date (the date of "death," the "last tumor measurement," "last date in drug log," or "last follow-up") was taken into consideration. The median duration of response with 95% CI was estimated using Kaplan Meier method.
Time Frame: Baseline up to PD or death (maximum up to 22 months)
Population: ITT population. The number of participants analyzed signifies the number of participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trastuzumab
Number analyzed (Participants) | 2
days | NA [NA to NA] — Data could not be estimated because disease progression was not documented.

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 6 month after last dose of study drug (maximum up to 22 months)
Population: Safety population included all participants who had received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
participants
  AEs | 4
  SAEs | 2

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Lab parameters assessed during the study were serum chemistry, biochemistry - serum electrolytes, hematology, 12 lead electrocardiogram, and urinalysis - protein, glucose, blood and other lab tests. Laboratory tests were graded according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) version 3.
Time Frame: Baseline up to 6 month after last dose of study drug (maximum up to 22 months)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
participants | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: The LVEF was measured using Multi Gated Acquisition (MUGA) or echocardiography (echocardiography was preferred), using the same technique throughout for consistency in an individual participant. Baseline LVEF assessments were done within 21 days prior to the start of treatment. Participants with clinically significant change from baseline (that is, absolute drop in LVEF of >=15%, and drop to a value <50%) have been reported.
Time Frame: Baseline, thereafter every 12 weeks (maximum up to 22 months)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
participants | 0

9. Secondary Outcome: Number of Participants With Human Epidermal Growth Factor Receptor 2 (HER2) Positive Gastric Cancer
Description: The HER2 status was determination by using immunohistochemistry (IHC) and confirmatory Fluorescent In Situ Hybridization (FISH) techniques. Only participants with HER2 positivity were allowed to receive study medication.
Time Frame: Baseline
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=4)
Anaemia (Blood and lymphatic system disorders) | 1
Deep vein thrombosis (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Melaena (Gastrointestinal disorders) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=4)
Diarrhoea (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Furuncle (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.